CLINICAL TRIAL: NCT06088940
Title: The Chemo-Gut Trial: A Double-blind Randomized Controlled Trial Investigating the Effects of a Multi-strain Probiotic on Gut Microbiota, Gastrointestinal Symptoms, and Psychosocial Health in Cancer Survivors
Brief Title: The Chemo-Gut Probiotic Trial for Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HREBA.CC-22-0289
Record Dates: First submitted 2023-05-18; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Psychosocial Problem; Gastrointestinal Dysfunction
Keywords: Gut microbiome; Patient Reported Outcomes; Probiotics; Cancer survivor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Theoretical Framework: This line of research follows the NIH ORBIT model for intervention development. Briefly, the ORBIT model provides a generic, systematic framework that emphasizes using a set of studies to form a chain of evidence that ultimately indicates readiness for an efficacy trial.
  Study Design. Consistent with the National Institutes for Health (NIH) clinical trial phases for drug development, this study will fit into phase II, where investigators are focused on examining treatment effectiveness. A placebo-controlled randomized double-blinded study design is the gold standard for intervention research involving medications or natural health products, such as probiotics.
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized individually upon enrollment after completing baseline assessments into the probiotic or placebo condition in a 1:1 allocation ratio using a computer-generated stratified randomization strategy (to balance age and sex). Randomization sequence will be pre-determined by randomization software and sequential allocations prepared in sealed envelopes, only to be revealed to a research assistant after consent and baseline questionnaires are completed. Once randomized, a research assistant will be responsible for assigning the probiotic or placebo for each participant to their study package so that the study coordinator, who will have direct contact with patients, will remain blinded to participants' condition. A member of the study team who does not have contact with participants will also be provided a copy of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Group 1: Experimental intervention) (Experimental): Participants will be given a 12-week supply of the probiotic supplement and asked to take 1 capsule daily by mouth at the same time as their first meal of the day.
  Interventions: Dietary Supplement: Multistrain Probiotic
- Placebo Group (Group 2: Control condition) (Placebo Comparator): Participants will be given a 12-week supply of the placebo capsules and asked to take 1 capsule daily by mouth at the same time as their first meal of the day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multistrain Probiotic — The probiotic capsule contains Lactobacillus and Bifidobacterium strains, ingested orally once daily.
  Arms: Probiotic Group (Group 1: Experimental intervention)
Other: Placebo — Placebo is composed of maltodextrin, that is an identically formulated and packaged inactive substance
  Arms: Placebo Group (Group 2: Control condition)

SUMMARY:
Purpose: The goal of this clinical trial is to determine whether probiotics can reduce gastrointestinal and psychosocial symptoms in post-treatment cancer survivors by impacting the gut microbiome.

Objectives: The main questions the investigators aim to answer are:

* Does taking the probiotic reduce gastrointestinal (e.g. belly pain) and psychosocial (e.g. depressive symptoms, fatigue) symptoms, and impact the gut microbiome?
* What relationships exist between gut bacteria, gastrointestinal, and psychosocial symptoms?

Methods: The study team will investigate this by giving a group of adult post-treatment cancer survivors either a probiotic capsule (intervention) or placebo capsule (control) over 12 weeks. Investigators will then analyze the bacterial diversity in participants' stool samples before and after these 12 weeks to see how the bacterial composition changed due to the treatment. Surveys will be used to ask participants questions about their physical and mental health, including specific gastrointestinal and psychosocial symptoms.

Implications: Cancer recovery is tough enough, and to minimize treatment-related long-term effects through a simple probiotic capsule would immensely improve the well-being and health of survivors.

DETAILED DESCRIPTION:
Background: Survivors of cancer experience chronic gastrointestinal (GI) and psychosocial health symptoms, and reduced gut microbial diversity. This may compromise survivors' long-term health and overall wellbeing. No studies have investigated probiotics for managing both GI and psychosocial symptoms together, or the composition of the gut microbiota in post-treatment cancer survivors.

Aims: To investigate the effects of a probiotic vs. placebo on (i) abdominal pain and depressive symptoms (primary outcomes); (ii) (a) GI (i.e. gas/bloating, diarrhea, constipation) and psychosocial (i.e. anxiety, cognitive function, fatigue) symptoms, and general health; and (b) gut microbiota composition; (iii) relationships between bacteria, GI and psychosocial symptoms.

Methods: This double-blinded, placebo-controlled, 2-arm, randomized trial will recruit N=66 participants allocated to the probiotic or placebo group for a 12-week trial. Adult survivors diagnosed with a solid tumour or blood cancer who have completed chemotherapy within the last 5 years, and show elevated GI or psychosocial symptoms will be included. The probiotic capsule contains Lactobacillus and Bifidobacterium strains, ingested orally once daily. Stool samples will be collected at baseline and week-12 and analyzed using GA-Map dysbiosis test and 16S rRNA gene sequencing. GI and psychosocial surveys will be completed at baseline, weeks 6 and 12. Descriptive statistics, frequencies, paired samples t-tests, linear mixed models, and Spearman's correlations analyses will be used.

Implications: This study explores a novel, microbiota-based treatment for chronic GI and psychosocial symptoms in cancer survivors. These findings and commitment to patient-centred knowledge translation via creating patient materials (e.g. infographics, personal results summary) will enable patients to make informed decisions about their health.

ELIGIBILITY:
Inclusion Criteria:

1. Male, female, and non-binary, any ethnicity
2. Aged 18 years or older
3. Diagnosed with hematological cancers (leukemia, Hodgkin's, and non-Hodgkin lymphoma), breast, osteosarcoma, Ewing's sarcoma, gynecological (cervical, endometrial), prostate, or testicular
4. Stages I - IV, including metastatic if stable and off treatment
5. Have received chemotherapy (with or without radiation, surgery, or hormone therapy)
6. Have completed primary cancer treatments
7. Within 5 years from their final cancer treatments, with emphasis placed on recruiting those within the first year post-treatment
8. Not currently pregnant or planning to become pregnant during the 12-week study
9. Evidence of clinically elevated levels (i.e. a score of 56 or higher) of GI and/or comorbid psychosocial symptoms as determined using PROMIS short forms for abdominal pain, gas/bloating, and general mental and physical health
10. Able to provide stool samples
11. Fluent in English, and have access to a computer, smartphone, or tablet with internet access to complete questionnaires
12. Provide written informed consent

Exclusion Criteria:

1. Diagnosis of central nervous system tumor, or colorectal cancer
2. Taken antibiotics and/or daily probiotic (including probiotic yogurt) within the 1 month prior to study participation
3. Currently or previously receiving immunotherapy
4. Diagnosed with irritable bowel syndrome or inflammatory bowel disease prior to being diagnosed with cancer
5. Diagnosed with a developmental/cognitive delay prior to cancer (e.g. autism spectrum disorder, downs syndrome)
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Effects of probiotic on abdominal pain | 12 weeks
  Endpoint: Clinically meaningful effects will be defined as reductions of 3 points or more from baseline scores of abdominal pain symptoms on PROMIS measures.
  Measure: PROMIS Belly Pain - Scale v1.0, 5a; Scores range from 20 to 80. Higher scores >60 indicate more symptoms.
Effects of probiotic on depression symptoms | 12 weeks
  Endpoint: Clinically meaningful effects will be defined as reductions of 3 points or more from baseline scores of depression on PROMIS measures.
  Measure: PROMIS Ca Item Bank v1.0 - Emotional Distress - Depression questionnaire; Scores range from 20 to 80. Higher scores >60 indicate more symptoms.

SECONDARY OUTCOMES:
Effects of probiotic on Gas/Bloating symptoms | 12 weeks
  Endpoint: Effects of probiotics on: Gas/bloating Measure: PROMIS Gas and Bloating - Scale v1.1 13a
Effects of probiotic on Diarrhea symptoms | 12 weeks
  Endpoint: Effects of probiotics on: Diarrhea Measure: PROMIS Diarrhea - Scale v1.0, 6a
Effects of probiotic on Constipation symptoms | 12 weeks
  Endpoint: Effects of probiotics on: Constipation Measure: PROMIS constipation - Scale v1.0, 9a
Effects of probiotic on anxiety symptoms | 12 weeks
  PROMIS Anxiety: v1.0 - Anxiety - Short Form 8a; Scores range from 20 to 80. Higher scores >60 indicate more symptoms.
Effects of probiotic on Fatigue symptoms | 12 weeks
  PROMIS v1.0 - Fatigue - Short Form 8a. Scores range from 20 to 80. Higher scores >60 indicate more symptoms.
Effects of probiotic on cognitive function | 12 weeks
  Measure: PROMIS v2.0 - Cognitive Function; Scores range from 80 (high function) to 20 (severe dysfunction).
Effects of probiotic on global health symptoms | 12 weeks
  Measure: PROMIS Global Health - Scale v1.2; Scores range from 80 (Excellent health) to 20 (Poor health).
Probiotic effects on gut microbiota alpha diversity composition | 12 weeks
  Measure: Chao1, Shannon, and Simpson index for statistically significant differences in alpha diversity between groups
Probiotic effects on gut microbiota beta diversity composition | 12 weeks
  Measure: Bray-Curtis index for statistically significant differences in beta diversity between groups
Probiotic effects on gut microbiota differential taxonomic abundance | 12 weeks
  Measure: statistically significant differences in differential taxonomic abundance (ASV's) between groups

OTHER OUTCOMES:
Relationships between bacterial taxa and symptoms | 12 weeks
  Measure: Scores for symptom outcomes will be correlated with bacterial operational taxonomic units (ASVs) using Spearman's rho for non-parametric data

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Deleemans, PhD, Study Director — University of Calgary Cumming School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published. Deidentified data will be made available to other researchers after primary data has been published and upon reasonable request to the PI.
Supporting Information: Study Protocol
Time Frame: 1. The study protocol is anticipated to be published by/before winter 2023
  2. Deidentified data will be made available to other researchers after primary data has been published (anticipated 2026)
Access Criteria: Reasonable request to the PI

REFERENCES:
- [Background] Deleemans JM, Chleilat F, Reimer RA, Henning JW, Baydoun M, Piedalue KA, McLennan A, Carlson LE. The chemo-gut study: investigating the long-term effects of chemotherapy on gut microbiota, metabolic, immune, psychological and cognitive parameters in young adult Cancer survivors; study protocol. BMC Cancer. 2019 Dec 23;19(1):1243. doi: 10.1186/s12885-019-6473-8. PMID 31870331
- [Background] Deleemans JM, Toivonen K, Reimer RA, Carlson LE. The Chemo-Gut Study: A Cross-Sectional Survey Exploring Physical, Mental, and Gastrointestinal Health Outcomes in Cancer Survivors. Glob Adv Health Med. 2022 Dec 21;11:2164957X221145940. doi: 10.1177/2164957X221145940. eCollection 2022. PMID 36583068
- [Background] Deleemans JM, Gajtani Z, Baydoun M, Reimer RA, Piedalue KA, Carlson LE. The Use of Prebiotic and Probiotic Interventions for Treating Gastrointestinal and Psychosocial Health Symptoms in Cancer Patients and Survivors: A Systematic Review. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211061733. doi: 10.1177/15347354211061733. PMID 34844479